CLINICAL TRIAL: NCT03951519
Title: Effect of Oral Water on the Quality of Volume Expansion in Resuscitation Patients: Pilot Study (The Water Study)
Brief Title: Effect of Oral Water on the Quality of Volume Expansion in Resuscitation Patients
Acronym: WATER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GUINOT 2018-2
Record Dates: First submitted 2019-05-10; First posted 2019-05-15 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Intubated-ventilated Patients in the Intensive Care Unit

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water (Experimental)
  Interventions: Other: oral administration of water
- Physiological serum (Active Comparator)
  Interventions: Other: administration of saline solution

INTERVENTIONS:
Other: oral administration of water — Volume expansion via 500 mL of water administered by the patient's nasogastric tube
  Arms: Water
Other: administration of saline solution — Volume expansion via 500 mL of saline (Nacl 0.9%) administered by the venous route
  Arms: Physiological serum

SUMMARY:
In ICU and operating theatre, fluid expansion is the main hemodynamic therapeutic. The objective of fluid expansion is to increase cardiac output thus arterial oxygen delivery to match patient's oxygen consumption. To date, it has been shown that all fluid expansion solutions may have side effects (hydro-electrolytic disorder, renal failure, hydro-sodium overload, etc.) that may limit their use.

Human digestive system physiologically ensures the absorption of oral water and hydration of the human body. Water is quickly absorbed by the digestive tract with a peak between 15 and 20 minutes. It has demonstrated that oral water remains the best hydration solution that have an effect on plasma volume expansion and cardiovascular system during exercise. While the cardiovascular effect of fluid expansion by saline serum is well known (venous return, preload and cardiac output), that of oral water vary in the literature depending on the physiological state of the patient and the clinical state. Oral water can change cardiac output and blood pressure through various physiological effects: increased blood volume, recruitment of splanchnic blood volume, and peripheral vasoconstriction. Usually, ICU patients have feeding through nasogastric tube.

To date, no study has studied the effect of a given amount of enteral cardiovascular system in ICU patients. The objective of this study is to describe the effect of oral water administration on the cardiovascular system of patients during the optimization and/or hemodynamic stabilization phase. The comparison of groups (water/ physiological saline) would allow us: (1) to describe the cardiovascular effects of water in the resuscitation patient, (2) to compare these cardiovascular effects with those of saline solution, (3) to have the data to design further study.

ELIGIBILITY:
Inclusion Criteria:

* Close family member has given written consent for patient included in emergency
* Intubated-ventilated patient in controlled volume mode
* Normothermal patient (36.5-37.5°C)
* Adult patient in intensive care for whom the attending physician has decided to give fluid expansion because of acute circulatory failure (systolic blood pressure < 90 mmHg, and/or mean blood pressure < 65 mmHg, and/or the need for infusion of vasopressor amines, and/or skin mottles, and/or diuresis < 0.5 mL/kg/h for a duration of ≥ 2 hours, and/or arterial lactate level > 2 mmol/L) (21),
* Patient with a variation OF SV over 10% with PLR,
* Echogenic patient,
* Patient with a regular sinus rhythm,
* Patient with a nasogastric tube.

Exclusion Criteria:

* Person subject to a legal protection measure (curatorship, guardianship)
* Person subject to a measure to safeguard justice
* Condition contraindicating the use of the oral route,
* Patient not affiliated or not covered by the national health system,
* Pregnant, parturient or breastfeeding woman,
* Hemodynamically unstable patient (variation of more than 10% in blood pressure),
* Arrhythmia-like rhythm disorder by atrial fibrillation,
* Modification of therapies (sedation, catecholamines) during the study period,
* Modification of the ventilatory parameters.
* Heart failure
* Oedemato-ascitic insufficiency of cirrhosis
* Changes in drug doses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
systolic ejection volume | 60 minutes
  variation in systolic ejection volume between base (time 1) and end of filling (time 2), expressed as a percentage.

SECONDARY OUTCOMES:
Blood pressure | immediately, 30 and 60 minutes after fluid administration
Cardiac output | immediately, 30 and 60 minutes after fluid administration,
volume of systolic ejections | immediately, 30 and 60 minutes after fluid administration
arterial lactate level | immediately after filling, 60 minutes after fluid administration,
Hourly diuresis | 60 minutes after fluid administration
change in DO2 | after filling, 60 minutes after fluid administration
change in VO2 | after filling, 60 minutes after fluid administration
number ofAdverse effects of water administration | "through study completion, an average of 1 year".
  (nausea, vomiting),
number Adverse effects of saline administration | "through study completion, an average of 1 year".
  (natremia, chloremia, acute pulmonary edema, renal failure).

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France

REFERENCES:
- [Result] Guinot PG, Nguyen M, Duclos V, Soudry-Faure A, Bouhemad B; Water Study Group. Oral water ingestion in the treatment of shock patients: a prospective randomized study. Intensive Care Med. 2020 Nov;46(11):2111-2112. doi: 10.1007/s00134-020-06215-y. Epub 2020 Aug 26. No abstract available. PMID 32851490
- [Derived] Guinot PG, Nguyen M, Duclos V, Berthoud V, Bouhemad B; water study group. Oral Water Has Cardiovascular Effects Up to 60 min in Shock Patients. Front Cardiovasc Med. 2021 Dec 20;8:803979. doi: 10.3389/fcvm.2021.803979. eCollection 2021. PMID 34988132